CLINICAL TRIAL: NCT05239806
Title: A Randomized, Double-blind Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01C (A Bivalent SARS-CoV-2 Trimeric Spike Protein Vaccine) and SCTV01E (A COVID-19 Alpha/Beta/Delta/Omicron Variants S-Trimer Vaccine) in Population Aged ≥12 Years Previously Fully Vaccinated With Inactivated COVID-19 Vaccine
Brief Title: A Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01C and SCTV01E in Population Aged ≥12 Years Previously Fully Vaccinated With Inactivated COVID-19 Vaccine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCTV01C/E-01-In-LAO-1
Record Dates: First submitted 2022-02-14; First posted 2022-02-15 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 infection; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCTV01C (Experimental): Participants will receive one dose of SCTV01C on Day 0 and one dose of SCTV01E on Day 180.
  Interventions: Biological: SCTV01C; Biological: SCTV01E
- SCTV01E (Experimental): Participants will receive one dose of SCTV01E on Day 0 and one dose of SCTV01E on Day 180.
  Interventions: Biological: SCTV01E
- Sinopharm inactivated COVID-19 vaccine (Active Comparator): Participants will receive one dose of Sinopharm inactivated COVID-19 vaccine on Day 0 and one dose of SCTV01E on Day 180.
  Interventions: Biological: Sinopharm inactivated COVID-19 vaccine; Biological: SCTV01E
- Comirnaty (Active Comparator): Participants will receive one dose of Comirnaty on Day 0 and one dose of SCTV01E on Day 180.
  Interventions: Biological: Comirnaty; Biological: SCTV01E

INTERVENTIONS:
Biological: SCTV01C — Day 0; intramuscular injection
  Arms: SCTV01C
Biological: SCTV01E — Day 0; intramuscular injection
  Arms: SCTV01E
Biological: Sinopharm inactivated COVID-19 vaccine — Day 0; intramuscular injection
  Arms: Sinopharm inactivated COVID-19 vaccine
Biological: Comirnaty — Day 0; intramuscular injection
  Arms: Comirnaty
Biological: SCTV01E — Day 180; intramuscular injection

SUMMARY:
The objective of study is to evaluate the immunogenicity and safety of SCTV01C or SCTV01E as booster compared with Sinopharm inactivated COVID-19 vaccine as booster. The study will also evaluate the immunogenicity and safety of 2-dose vaccinations.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, and approved vaccine-controlled Phase II booster study. It will evaluate the immunogenicity and safety of one dose of SCTV01C or SCTV01E as booster compared with one dose of Sinopharm inactivated COVID-19 vaccine or one dose of Commirnaty as booster. The study will also evaluate the immunogenicity and safety of 2-dose vaccinations (1-dose of SCTV01C and 1-dose of SCTV01E, or 2-dose of SCTV01E, or 1-dose of Sinopharm inactivated COVID-19 vaccine and 1-dose of SCTV01E, 1-dose of Comirnaty and 1-dose of SCTV01E).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥12 years old when signing ICF;
2. Participants who were fully vaccinated with inactivated COVID-19 vaccine (Sinopharm inactivated COVID-19 vaccine), and the interval between the last dose and this study vaccination is ≥3 months and ≤12 months;
3. The participant and/or his legal guardian and/or his entrusted person can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. The participant and/or his legal guardian and/or his entrusted person have the ability to read, understand, and fill in record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the 1st study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

1. Previously diagnosed with COVID-19;
2. Presence of fever within 3 days before the study vaccination;
3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or other disease corresponding use of immunosuppressants;
4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (except for skin basal cell carcinoma and carcinoma in-situ of cervix), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants received other drugs or vaccines used to prevent COVID-19 (exception for Sinopharm inactivated COVID-19 vaccine) ;
15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
17. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
18. Those who plan to donate ovum or sperms during the study period;
19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
21. Those who are tested positive for HIV in terms of serology.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
GMT of neutralizing antibodies against Delta (B.1.617.2) variant on Day 28. | Day 28 after the study vaccination
GMT of neutralizing antibodies against Omicron (B.1.1.529) variant on Day 28. | Day 28 after the study vaccination
GMT of neutralizing antibodies against Delta (B.1.617.2) variant on Day 208. | Day 208 after the study vaccination
GMT of neutralizing antibodies against Omicron (B.1.1.529) variant on Day 208. | Day 208 after the study vaccination

SECONDARY OUTCOMES:
Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subsets on Day 28 and Day 208. | Day 28 and D208 after the study vaccination
Seroresponse rates of neutralizing antibodiesto Delta variant on Day 28. | Day 28 after the study vaccination
Seroresponse rates of neutralizing antibodies to Omicron variant rates on Day 28. | Day 28 after the study vaccination
Seroresponse rates of neutralizing antibodies to Delta variant on Day 208. | Day 208 after the study vaccination
Seroresponse rates of neutralizing antibodies to Omicron variant on Day 208. | Day 208 after the study vaccination
Incidence and severity of solicited AEs of SCTV01C from Day 0 to Day 7 and Day 180 to Day 187. | Day 0 to Day 7 after the 1st study vaccination and Day 180 to Day 187 after the 2nd study vaccination
Incidence and severity of all unsolicited AEs of SCTV01C from Day 0 to Day 28 and Day 180 to Day 208. | Day 0 to Day 28 after the 1st study vaccination and Day 180 to Day 208 after the 2nd study vaccination
Incidence and severity of SAEs and AESIs of SCTV01C within 365 days. | Day 0 to Day 365 after the 1st study vaccination
Incidence and severity of solicited AEs of SCTV01E from Day 0 to Day 7 and Day 180 to Day 187. | Day 0 to Day 7 after the 1st study vaccination and Day 180 to Day 187 after the 2nd study vaccination
Incidence and severity of all unsolicited AEs of SCTV01E from Day 0 to Day 28 and Day 180 to Day 208. | Day 0 to Day 28 after the 1st study vaccination and Day 180 to Day 208 after the 2nd study vaccination
Incidence and severity of SAEs and AESIs of SCTV01E within 365 days. | Day 0 to Day 365 after the 1st study vaccination